CLINICAL TRIAL: NCT01974206
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial to Evaluate the Efficacy and Safety of a Vaccine, ASP0113, in Cytomegalovirus (CMV)-Seronegative Kidney Transplant Recipients Receiving an Organ From a CMV-Seropositive Donor
Brief Title: A Study to Evaluate the Efficacy and Safety of a Vaccine, ASP0113, in Cytomegalovirus (CMV)-Seronegative Kidney Transplant Recipients Receiving an Organ From a CMV-Seropositive Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Vical (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0113-CL-2001; 2013-000464-29 (EudraCT Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation Cytomegalovirus (CMV) Negative Recipients
Keywords: ASP0113; Cytomegalovirus (CMV); Kidney Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP0113 (Experimental): Participants received 1 mL of 5 mg/mL of ASP0113 via injection in the deltoid muscle alternating sides with each dose on days 30, 60, 90, 120 and 180 in relation to the day of transplant (Day 0).
  Interventions: Biological: ASP0113
- Placebo (Placebo Comparator): Participants received 1 mL of 5 mg/mL of placebo via injection in the deltoid muscle alternating sides with each dose on days 30, 60, 90, 120 and 180 in relation to the day of transplant (Day 0).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ASP0113 — intramuscular injection
  Arms: ASP0113
Drug: Placebo — intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy of ASP0113 compared to placebo in reducing the incidence of cytomegalovirus (CMV) viremia in CMV-seronegative subjects receiving a kidney from a CMV-seropositive donor. This study also evaluated the safety of ASP0113 in this patient population.

DETAILED DESCRIPTION:
Participants were followed for one year after first study drug injection. This was the primary study period.

Participants were followed for 4.5 years after completion of the primary study to assess long-term safety of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* CMV negative subject having received a CMV seropositive kidney (living or deceased)
* Participant started valganciclovir or ganciclovir within 10 days of transplant and had received it through Randomization.

Exclusion Criteria:

* Participant underwent a course of CMV-specific prophylactic therapy with antiviral drugs with a duration of greater than 100 days.
* Participant had received from one month prior to transplant or planned to receive CMV immunoglobulin.
* Participant had CMV viremia or CMV disease from time of transplant until time of Randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (53):
- United States (33):
  - Site US10026, Phoenix, Arizona
  - Site US10003, Los Angeles, California
  - Site US10004, San Diego, California
  - Site US10036, San Francisco, California
  - Site US10037, San Francisco, California
  - Site US10044, Aurora, Colorado
  - Site US10018, New Haven, Connecticut
  - Site US10058, Atlanta, Georgia
  - Site US10013, Atlanta, Georgia
  - Site US10030, Chicago, Illinois
  - Site US10009, Chicago, Illinois
  - Site US10057, Indianapolis, Indiana
  - Site US10046, Lexington, Kentucky
  - Site US10041, New Orleans, Louisiana
  - Site US10049, Portland, Maine
  - Site US10023, Ann Arbor, Michigan
  - Site US10048, Detroit, Michigan
  - Site US10016, St Louis, Missouri
  - Site US10015, Omaha, Nebraska
  - Site US10045, Buffalo, New York
  - Site US10012, The Bronx, New York
  - Site US10050, Greenville, North Carolina
  - Site US10001, Cleveland, Ohio
  - Site US10042, Pittsburgh, Pennsylvania
  - Site US10047, Charleston, South Carolina
  - Site US10027, Nashville, Tennessee
  - Site US10028, Houston, Texas
  - Site US10014, Salt Lake City, Utah
  - Site US10038, Charlottesville, Virginia
  - Site US10031, Richmond, Virginia
  - Site US10020, Seattle, Washington
  - Site US10011, Seattle, Washington
  - Site US10029, Madison, Wisconsin
- Australia (3):
  - Site AU61002, Sydney, New South Wales
  - Site AU61004, Woolloongabba, Queensland
  - Site AU61001, Adelaide SA, South Australia
- Canada (4):
  - Site CA15004, Vancouver, British Columbia
  - Site CA15003, Halifax, Nova Scotia
  - Site CA15005, London, Ontario
  - Site CA15006, Toronto, Ontario
- France (4):
  - Site FR33005, Bordeaux
  - Site FR33003, Montpellier
  - Site FR33004, Nantes
  - Site FR33001, Nice
- Germany (5):
  - Site DE49002, Berlin
  - Site DE49001, Berlin
  - Site DE49008, Bonn
  - Site DE49003, Erlangen
  - Site DE49005, Hamburg
- Spain (4):
  - Site ES34003, Barcelona
  - Site ES34002, Barcelona
  - Site ES34001, Barcelona
  - Site ES34004, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Vincenti F, Budde K, Merville P, Shihab F, Ram Peddi V, Shah M, Wyburn K, Cassuto-Viguier E, Weidemann A, Lee M, Flegel T, Erdman J, Wang X, Lademacher C. A randomized, phase 2 study of ASP0113, a DNA-based vaccine, for the prevention of CMV in CMV-seronegative kidney transplant recipients receiving a kidney from a CMV-seropositive donor. Am J Transplant. 2018 Dec;18(12):2945-2954. doi: 10.1111/ajt.14925. Epub 2018 Jun 20. PMID 29745007
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=0113-CL-2001
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14616&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 150 participants were enrolled into the study from 6 countries. Eligible participants were ≥18 years of age, CMV-seronegative at the time of the transplant and had a kidney allograft from a CMV-seropositive living or deceased donor. After the primary period completion, 149 participants entered the long-term follow-up period.
Pre-assignment Details: Screening assessments were performed from 14-30 days after the transplant. Participants were randomized at day 30 in relation to the day of the transplant, in a 1:1 ratio to ASP0113 or placebo. Participants were stratified by the use of antithymocyte globulin (ATG) prior to randomization and by the receipt of a kidney from a living or deceased donor.
Groups:
- ASP0113 5mg: Participants received 1 mL of 5 mg/mL of ASP0113 via injection in the deltoid muscle alternating sides with each dose on days 30, 60, 90, 120 and 180 in relation to the day of transplant (Day 0).
Period: Overall Study
Arm/Group | Placebo | ASP0113 5mg
Started | 74 | 76
Received Treatment | 74 | 75
Completed | 68 | 75
Not Completed | 6 | 1
Not completed — Did Not Take Study Drug | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population: Age, Gender, Race, Ethnicity Randomized population: Use of ATG, Source of current Transplant, randomization strata
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ASP0113 | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (13.3) | 50.8 (13.6) | 49.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 55 | 55 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 70 | 72
  Not Hispanic or Latino | 72 | 6 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 57 | 61 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Use of ATG [Count of Participants; unit: Participants]
  No | 44 | 44 | 88
  Yes | 30 | 32 | 62
Randomization Strata [Count of Participants; unit: Participants]
  Living Donor & ATG Use = No | 18 | 16 | 34
  Living Donor & ATG Use = Yes | 8 | 10 | 18
  Deceased Donor & ATG Use = Yes | 22 | 22 | 44
  Deceased Donor & ATG Use = No | 26 | 27 | 53
  Not Recorded | 0 | 1 | 1
Source of Current Transplant [Count of Participants; unit: Participants]
  LIVING UNRELATED DONOR | 10 | 17 | 27
  LIVING RELATED DONOR | 16 | 9 | 25
  DECEASED DONOR | 48 | 49 | 97
  Not Recorded | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With CMV Viremia Through 1 Year Post First Study Drug Injection
Description: CMV viremia was defined as presence of cytomegalovirus as measured in plasma viral load of ≥ 1000 IU/mL by central laboratory assay. A participant who discontinued the study without a positive CMV viral load was imputed as having a CMV viremia. A participant who had more than one viral load ≥ 1000 IU/mL by central assay was counted once in this summary. CMV viral loads after first injection (Day 1) through Day 380 (scheduled or unscheduled) were included in the analysis.
Time Frame: From first study dose injection (day 1) up to one year post study drug injection (up to Day 380)
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least 1 dose of randomized study drug and who had at least 1 post dose viral load assessment within 1 year post first injection by central laboratory.
Measure: Number; unit: Percentage of Paticipants
Arm/Group | Placebo | ASP0113 5mg
Number analyzed (Participants) | 73 | 73
Percentage of Paticipants
  Known CMV viremia | 35.6 | 35.6
  Imputed CMV viremia due to discontinuation | 5.5 | 0
Statistical Analysis 1: Comparison: Placebo vs ASP0113 5mg; The Cochran-Mantel-Haenszel (CMH) estimate of the common odds ratio (ASP0113 vs placebo) stratified by randomization strata, and the 90% CIs of the CMH odds ratio stratified by randomization group; Test type: Other; p = 0.307, Cochran-Mantel-Haenszel — P-value (1-sided) of the Exact Cochran-Mantel-Haenszel method adjusted odds ratio stratified by randomization group; Common Odds Ratio = 0.79, 90% CI 2-sided [0.43 to 1.47]

2. Secondary Outcome: Percentage of Participants With Adjudicated CMV-Associated Disease, Including CMV Syndrome and CMV Tissue-Invasive Disease (Primary Study Period)
Description: An independent panel of medical experts reviewed/adjudicated events of CMV-associated disease including CMV syndrome and tissue invasive disease, which were defined according to the American Society of Transplantation Recommendations for Screening, Monitoring and Reporting of Infectious Complications in Immunosuppression Trials in Recipients of Organ Transplantation 2006.
Time Frame: From first study dose injection (day 1) up to one (up to Day 380) year post study drug injection
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113 5mg
Number analyzed (Participants) | 73 | 73
Percentage of Participants | 19.18 | 19.18
Statistical Analysis 1: Comparison: Placebo vs ASP0113 5mg; The exact Cochran-Mantel-Haenszel (CMH) estimate of the common odds ratio (ASP0113 vs placebo) stratified by randomization group, and the 90% CI of the exact CMH odds ratio stratified by randomization group; Test type: Other; p = 0.576, Cochran-Mantel-Haenszel — P-value (1-sided) of the Exact Cochran-Mantel-Haenszel method adjusted odds ratio stratified by randomization group; Common Odds Ratio = 0.99, 90% CI 2-sided [0.46 to 2.15]

3. Secondary Outcome: Percentage of Participants With Plasma Viral Load ≥ The Lower Limit of Quantification (LLOQ) Assessed by Central Laboratory (Primary Study Period)
Description: The central laboratory had the LLOQ level for CMV viral load assessment. When the viral load was below the LLOQ the actual reading was not possible and was denoted as ≤LLOQ. If the participant had any CMV viral load assessments greater than the LLOQ, set up by the central laboratory, participant was classified as viremic and was included in the analysis.
Time Frame: From first study dose injection (day 1) up to one year post study drug injection (up to Day 380)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113 5mg
Number analyzed (Participants) | 73 | 73
Percentage of Participants | 49.32 | 46.58
Statistical Analysis 1: Comparison: Placebo vs ASP0113 5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.408, Cochran-Mantel-Haenszel — P-value (1-sided) of the Exact Cochran-Mantel-Haenszel method adjusted odds ratio stratified by randomization group; Common Odds Ratio = 0.88, 90% CI 2-sided [0.48 to 1.59]

4. Secondary Outcome: Percentage of Participants Who Took Adjudicated CMV-specific Antiviral Therapy for the Treatment of CMV Viremia or Disease (Primary Study Period)
Description: An independent panel of medical experts reviewed/adjudicated events of CMV-specific AVT for treatment of CMV viremia or disease.
Time Frame: From first study dose injection (day 1) up to one year post study drug injection (up to Day 380)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113 5mg
Number analyzed (Participants) | 73 | 73
Percentage of Participants | 45.21 | 42.47
Statistical Analysis 1: Comparison: Placebo vs ASP0113 5mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.419, Cochran-Mantel-Haenszel — P-value (1-sided) of the Exact Cochran-Mantel-Haenszel method adjusted odds ratio stratified by randomization group; Common Odds Ratio = 0.88, 90% CI 2-sided [0.48 to 1.61]

5. Secondary Outcome: Percentage of Participants With Graft Survival (Primary Study Period)
Description: Graft survival was defined for any participant that did not fit the definition of graft loss. Graft loss was defined as participant death, re-transplant, nephrectomy, or return to permanent dialysis (i.e., for > 30 days). Missing values for graft survival were not included in the denominator when making the proportion. The analysis population was the FAS.
Time Frame: From first study dose injection (day 1) up to one year post study drug injection (up to Day 380)
Population: The analysis population was the FAS, with data available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113 5mg
Number analyzed (Participants) | 68 | 71
Percentage of Participants | 98.53 | 100
Statistical Analysis 1: Comparison: Placebo vs ASP0113 5mg; Exact Cochran-Mantel-Haenszel estimate of the common odds ratio could not be calculated as 100% of ASP0113 group showed graft survival, and this leads to having a value of 0 for the denominator for the ratio thus odds ratio is not estimable. The 90% CI (2-sided) values for the odds ratio are 0.11 to NA, where NA is an infinity value; Test type: Other; p = 0.5, Cochran-Mantel-Haenszel — P-value (1-sided) of the Exact Cochran-Mantel-Haenszel method adjusted odds ratio stratified by randomization group

6. Secondary Outcome: Percentage of Participants With Graft Survival (Long-term Follow up)
Description: Graft survival was defined for any participant that did not fit the definition of graft loss. Graft loss was defined as participant death, re-transplant, nephrectomy, or return to permanent dialysis (i.e., for > 30 days). Missing values for graft survival were not included in the denominator when making the proportion.
Time Frame: Month 18, 30, 42, 54, and 66
Population: All participants who entered long-term follow-up.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | ASP0113 5mg
Number analyzed (Participants) | 74 | 76
Percentage of Participants
  Long Term Follow Up Month 18 | 91.9 | 94.7
  Long Term Follow Up Month 30 | 83.8 | 81.6
  Long Term Follow Up Month 42 | 85.1 | 80.3
  Long Term Follow Up Month 54 | 78.4 | 77.6
  Long Term Follow Up Month 66 | 82.4 | 84.2

ADVERSE EVENTS:
Time Frame: Day 1 to Day 380
Description: Treatment Emergent Adverse Event (TEAE) was defined as an adverse event observed after the first study drug injection Day 1 through Day 380. No AEs were collected / reported during the long-term follow-up period.
Arm/Group | Placebo | ASP0113
All-Cause Mortality (participants affected / at risk) | 5/74 | 7/75
Serious Adverse Events (participants affected / at risk) | 36/74 | 44/75
Other Adverse Events (participants affected / at risk) | 72/74 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=74) | ASP0113 (N=75)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Hyperparathyroidism tertiary (Endocrine disorders) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (3) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 4 (4) | 3 (3)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 0 (0) | 2 (3)
Bacterial pyelonephritis (Infections and infestations) | 1 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 7 (7)
Cytomegalovirus mucocutaneous ulcer (Infections and infestations) | 0 (0) | 1 (2)
Cytomegalovirus oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus syndrome (Infections and infestations) | 5 (5) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 3 (3) | 5 (7)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Epstein-Barr viraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 5 (6)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Polyomavirus-associated nephropathy (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (4)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 3 (4)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Perinephric collection (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 5 (5)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
HLA marker study positive (Investigations) | 0 (0) | 1 (1)
Immunosuppressant drug level increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 6 (10) | 10 (12)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder atrophy (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Ureteral stent removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Urostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=74) | ASP0113 (N=75)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 19 (23) | 29 (32)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) | 10 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 5 (5)
Tachycardia (Cardiac disorders) | 3 (3) | 5 (5)
Vision blurred (Eye disorders) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 6 (7) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 24 (38) | 23 (33)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (19) | 13 (22)
Vomiting (Gastrointestinal disorders) | 9 (13) | 9 (12)
Asthenia (General disorders) | 8 (8) | 5 (5)
Chills (General disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 24 (38) | 27 (59)
Injection site erythema (General disorders) | 2 (2) | 8 (14)
Injection site pain (General disorders) | 18 (46) | 47 (277)
Oedema (General disorders) | 3 (3) | 5 (5)
Oedema peripheral (General disorders) | 5 (8) | 9 (13)
Pyrexia (General disorders) | 13 (14) | 9 (11)
BK virus infection (Infections and infestations) | 16 (18) | 16 (17)
Cytomegalovirus infection (Infections and infestations) | 5 (7) | 3 (4)
Cytomegalovirus syndrome (Infections and infestations) | 6 (6) | 7 (7)
Cytomegalovirus viraemia (Infections and infestations) | 19 (22) | 22 (30)
Escherichia urinary tract infection (Infections and infestations) | 5 (5) | 6 (9)
Nasopharyngitis (Infections and infestations) | 8 (10) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 8 (9)
Urinary tract infection (Infections and infestations) | 4 (5) | 10 (17)
Urinary tract infection bacterial (Infections and infestations) | 3 (5) | 8 (11)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 6 (10)
Blood creatinine increased (Investigations) | 16 (19) | 11 (17)
Weight increased (Investigations) | 3 (3) | 4 (4)
White blood cell count decreased (Investigations) | 4 (12) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (8) | 12 (16)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 5 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (8) | 7 (8)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (4) | 11 (12)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (22) | 21 (38)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (5)
Dizziness (Nervous system disorders) | 9 (12) | 3 (3)
Headache (Nervous system disorders) | 12 (14) | 13 (13)
Tremor (Nervous system disorders) | 7 (9) | 10 (11)
Insomnia (Psychiatric disorders) | 6 (8) | 8 (11)
Dysuria (Renal and urinary disorders) | 6 (6) | 5 (5)
Haematuria (Renal and urinary disorders) | 7 (7) | 6 (8)
Kidney fibrosis (Renal and urinary disorders) | 4 (4) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Ureteral stent removal (Surgical and medical procedures) | 6 (6) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 9 (14) | 12 (12)
Hypotension (Vascular disorders) | 8 (10) | 11 (16)
Orthostatic hypotension (Vascular disorders) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2014-01-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT01974206/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT01974206/SAP_001.pdf